CLINICAL TRIAL: NCT05327660
Title: Remote Carbon Monoxide Monitoring and Incentives for Tobacco Cessation in Quitlines
Brief Title: CO Monitoring for Tobacco Cessation in Quitlines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Consumer Wellness Solutions (Industry)
Collaborators: Vincere Health (Industry); Maryland State Tobacco Quitline (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-0056
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Tobacco Dependence
Keywords: tobacco cessation; tobacco quitlines; carbon monoxide monitoring; incentives
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Quitline treatment as usual (TAU) (Active Comparator): Quitline services provided by participating state quitlines
  Interventions: Combination Product: Quitline Treatment as Usual (TAU)
- Quitline TAU plus remote CO monitoring (Experimental): Quitline service plus daily CO monitoring via a smartphone app
  Interventions: Combination Product: Quitline Treatment as Usual (TAU); Combination Product: Remote Carbon Monoxide (CO) Monitoring
- Quitline TAU plus incentivized remote CO monitoring (Experimental): Quitline TAU plus remote CO monitoring with small monetary incentives
  Interventions: Combination Product: Quitline Treatment as Usual (TAU); Combination Product: Incentivized Remote CO Monitoring

INTERVENTIONS:
Combination Product: Quitline Treatment as Usual (TAU) — Quitline TAU is services provided by the state quitline and includes phone coaching, nicotine replacement, supplemental materials (e.g., text messaging, online content).
Combination Product: Remote Carbon Monoxide (CO) Monitoring — Remote CO monitoring includes a smartphone app and a remote carbon monoxide monitor. The app tracks and prompts daily use of the CO monitor.
  Arms: Quitline TAU plus remote CO monitoring
Combination Product: Incentivized Remote CO Monitoring — Incentivized remote CO monitoring includes a smartphone app and a remote carbon monoxide monitor. The app tracks and prompts daily use of the CO monitor and delivers small monetary incentives for each use of the CO monitor.
  Arms: Quitline TAU plus incentivized remote CO monitoring

SUMMARY:
The present study is a 3-arm randomized controlled pilot study. Participants who call the Maryland Tobacco Quitline and are eligible for study participation are randomized to receive quitline tobacco cessation treatment as usual (TAU), TAU plus remote carbon monoxide (CO) monitoring via smartphone app, or TAU plus remote carbon monoxide monitoring plus incentives vis smartphone app. The investigators hypothesize that remote CO monitoring will be feasible and acceptable to deliver in the quitline setting, will increase treatment engagement, and will increase tobacco cessation and treatment satisfaction rates.

ELIGIBILITY:
Inclusion Criteria:

* Daily cigarette smokers calling into participating quitlines
* 18 year or older
* Reads and speaks English
* Has a smartphone with a data plan
* Willing to download and use study app
* Willing to use CO monitor

Exclusion Criteria:

• Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Carpenter, PhD, Principal Investigator — Consumer Wellness Solutions
Locations (1):
- Optum Center for Wellbeing Research, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring
Started | 73 | 76 | 80
Completed | 73 | 76 | 80
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring | Total
Number analyzed (Participants) | 73 | 76 | 80 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (11.8) | 54.5 (11.7) | 55.5 (11.1) | 54.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 49 | 48 | 143
  Male | 27 | 27 | 32 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5 | 10
  Not Hispanic or Latino | 69 | 72 | 71 | 212
  Unknown or Not Reported | 2 | 1 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 4
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 30 | 42 | 35 | 107
  White | 32 | 30 | 36 | 98
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 73 | 76 | 80 | 229

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction
Description: Rating of satisfaction with quitline services on a 6-point scale collected via follow-up survey. Five questions were internally developed to determine satisfaction with the quitline services provided where low numbers (1-3) mean dissatisfaction and high numbers (4-6) mean satisfaction. Participants that reported a score of 4 (somewhat satisfied) or more are represented in the data table.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring
Number analyzed (Participants) | 41 | 47 | 59
Participants | 38 | 44 | 56

2. Primary Outcome: Treatment Engagement
Description: Number of quitline calls each participant engages in, collected via clinical record system.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: Calls completed
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring
Number analyzed (Participants) | 73 | 76 | 80
Calls completed | 2.2 (1.4) | 2.3 (1.6) | 2.7 (1.9)

3. Primary Outcome: Self-reported Tobacco Abstinence
Description: 7 day point prevalence abstinence from all combustible tobacco collected via follow-up survey
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring
Number analyzed (Participants) | 73 | 76 | 80
Participants | 15 | 18 | 25

4. Secondary Outcome: Biochemically Verified Tobacco Abstinence
Description: CO monitor reading 60 days post randomization (must be 7ppm or less to be considered abstinent) collected via smartphone app
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring
Number analyzed (Participants) | 73 | 76 | 80
Participants | 6 | 14 | 20

5. Secondary Outcome: Engagement With CO Monitor
Description: Number of times remote CO monitor is used collected via smartphone app.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: Breath tests completed
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring
Number analyzed (Participants) | 26 | 55 | 56
Breath tests completed | 7.7 (7.3) | 54.8 (49.6) | 80.9 (48.5)

6. Secondary Outcome: Satisfaction With CO Monitor
Description: Satisfaction with CO monitor measures on a 6-point scale collected via follow-up survey. Five questions were internally developed to determine satisfaction with the CO monitor device and app where low numbers (1-3) mean dissatisfaction and high numbers (4-6) mean satisfaction. Participants that reported a score of 4 (somewhat satisfied) or more are represented in the data table.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring
Number analyzed (Participants) | 34 | 42 | 55
Participants | 30 | 38 | 51

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 8 months, from the start of recruitment through the final outcome survey collection.
Arm/Group | Quitline Treatment as Usual (TAU) | Quitline TAU Plus Remote CO Monitoring | Quitline TAU Plus Incentivized Remote CO Monitoring
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/76 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/76 | 0/80
Other Adverse Events (participants affected / at risk) | 0/73 | 0/76 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT05327660/Prot_SAP_000.pdf